CLINICAL TRIAL: NCT01256463
Title: HIV Prevention for People Living With HIV/AIDS: Evaluation of an Intervention Toolkit for HIV Care and Treatment Settings
Brief Title: HIV Prevention for PLHIV: Evaluation of an Intervention Toolkit for HIV Care & Treatment Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Columbia University (Other); Ministry of Health and Social Services, Namibia (Other Government); Kenya Ministry of Health (Other Government); Ministry of Health, Tanzania (Other Government); Ministry of Health and Social Welfare, Zanzibar (Other Government)
Responsible Party: Principal Investigator, Daniel Kidder, Health Scientist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-CGH-5540
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison (No Intervention)
- HIV prevention intervention (Experimental): The HIV prevention intervention will be delivered to HIV-seropositive patients in HIV care and treatment clinics during all routine visits. Health care providers (including physicians, clinical officers, and nurses) will deliver HIV prevention messages on correct and consistent condom use, disclosure of serostatus, partner HIV testing, adherence and alcohol reduction during clinic visits. Health care providers will also assess and treat sexually transmitted infections (STIs), and provide basic contraceptives and brief safer pregnancy counseling.
  Interventions: Behavioral: HIV prevention intervention

INTERVENTIONS:
Behavioral: HIV prevention intervention
  Arms: HIV prevention intervention

SUMMARY:
The rapid scale-up of HIV care and treatment in resource-limited settings provides the opportunity to reach many HIV-positive individuals with prevention messages and interventions in care and treatment settings. However, HIV prevention is rarely incorporated into the routine care and treatment of people living with HIV, leaving missed opportunities to reach patients with critical interventions.

This study will evaluate an HIV prevention intervention package for health care settings in sub-Saharan Africa. The HIV prevention intervention will be delivered to HIV-seropositive patients in HIV care and treatment clinics during all routine visits. Health care providers (HCPs) will deliver HIV prevention messages on correct and consistent condom use, disclosure of serostatus, partner HIV testing, adherence and alcohol reduction. They will also assess and treat sexually transmitted infections (STIs) and provide basic contraceptives and safer pregnancy counseling.

Trained lay counselors (LCs) will deliver HIV prevention interventions in the clinics. LCs will be persons without medical training, many of whom will be PLHIV, who will be trained to provide HIV prevention counseling, promote HIV testing of partners and children (and provide HIV testing where allowed by national guidelines), and counsel HIV-positive patients on medication adherence and alcohol use.

The prevention intervention package will be evaluated in HIV clinics in three sub-Saharan African countries: Kenya, Namibia, and Tanzania. This project will be a longitudinal group-randomized trial with 9 intervention clinics (3 per country) and 9 comparison clinics (3 per country). Two hundred patients per clinic (total N = 3600) will be followed for 12 months. This evaluation will examine the effectiveness of the HIV prevention interventions delivered by HCPs and LCs on patient-level outcomes such as risky sexual behavior, disclosure of HIV status, partner HIV testing, alcohol use, HIV antiretroviral (ARV) medication adherence, STI treatment, pregnancies, and contraceptive use.

In addition to the patient outcomes, the acceptability of the interventions and materials, as well as the feasibility of integrating the interventions into HIV care and treatment settings, will be assessed.

Data will be collected via patient interviews, HCP and LC questionnaires, observations of HCP and LC patient visits, patient medical chart review, and review of clinic service data.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* HIV-positive patients receiving care at a project clinic and seen at the clinic at least twice prior to enrollment
* Sexually active within the past three months
* Planning to attend the clinic for at least 1 year
* Able to conduct interview in one of the following languages:

Kenya: English, Kiswahili Namibia: English, Oshiwambo, Damara-nama, Otjiherero, Afrikaans Tanzania: English, Kiswahili

* Able to provide informed consent to participate in the project

Exclusion Criteria:

* Younger than 18 years of age
* Not sexually active within the last three months
* Planning to move from the vicinity of the clinic within one year
* Not enrolled in the HIV clinic and/or have not been seen for at least two clinic visits
* Cannot provide informed consent
* Patients who are acutely ill or are determined by clinical staff to be too ill to participate
* Spouses or identified partners of participating patients
* Pregnant women and male partners of pregnant women, as family planning counseling and unintended pregnancy are some of the primary study outcomes
* Not able to complete interview in one of the languages in the inclusion criteria
* Participated in pilot study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3548 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Unprotected vaginal and anal sex | Baseline
Unprotected vaginal and anal sex | 6 month follow-up
Unprotected vaginal and anal sex | 12-month follow-up

SECONDARY OUTCOMES:
Number of sex partners | Baseline
Number of sex partners | 6 month follow-up
Number of sex partners | 12 month follow-up
Number of sex partners getting an HIV test | Baseline
Number of sex partners getting an HIV test | 6 month follow-up
Number of sex partners getting an HIV test | 12 month follow-up
Disclosure of HIV status to sex partners | Baseline
Disclosure of HIV status to sex partners | 6 month follow-up
Disclosure of HIV status to sex partners | 12-month follow-up
Alcohol use | Baseline
Alcohol use | 6 month follow-up
Alcohol use | 12-month follow-up
Adherence to HIV antiretroviral medications | Baseline
Adherence to HIV antiretroviral medications | 6 month follow-up
Adherence to HIV antiretroviral medications | 12-month follow-up
Unintended pregnancy or partner pregnancy | Baseline
Unintended pregnancy or partner pregnancy | 6 month follow-up
Unintended pregnancy or partner pregnancy | 12-month follow-up
Provision of family planning counseling and services | Baseline
Provision of family planning counseling and services | 6 month follow-up
Provision of family planning counseling and services | 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Bachanas, PhD, Principal Investigator — Centers for Disease Control and Prevention; Daniel Kidder, PhD, Study Director — Centers for Disease Control and Prevention

REFERENCES:
- [Derived] Kidder DP, Bachanas P, Medley A, Pals S, Nuwagaba-Biribonwoha H, Ackers M, Howard A, Deluca N, Mbatia R, Sheriff M, Arthur G, Katuta F, Cherutich P, Somi G; PwP Evaluation Study team. HIV prevention in care and treatment settings: baseline risk behaviors among HIV patients in Kenya, Namibia, and Tanzania. PLoS One. 2013;8(2):e57215. doi: 10.1371/journal.pone.0057215. Epub 2013 Feb 25. PMID 23459196